CLINICAL TRIAL: NCT06885203
Title: Social and Environmental Determinants of Breast Cancer Survivorship: the Black Breast Cancer Survivor's Intervention (BBCSI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1563; NCI-2025-02122 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-03-18; First posted 2025-03-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Participants will be recruited through our Community Based Organizations (CBOs) and other community collaborator networks.
  Interventions: Behavioral: Black Breast Cancer Survivor's Intervention
- Wait-List (start in week 7) (Experimental): Participants will be recruited through our Community Based Organizations (CBOs) and other community collaborator networks.
  Interventions: Behavioral: Black Breast Cancer Survivor's Intervention

INTERVENTIONS:
Behavioral: Black Breast Cancer Survivor's Intervention — Participants will complete the BBCSI course (1-hour virtual sessions every week for 6 weeks), answer questionnaires before and after the course, and provide urine samples.

SUMMARY:
The goal of this research study is to learn about the effects of the BBCSI course on the quality of life of Black breast cancer survivors.

A community-based and peer-led Black Breast Cancer Survivor's Intervention (BBCSI) course has been developed to help improve the quality of life of Black breast cancer survivors.

DETAILED DESCRIPTION:
Primary Objectives:

Guided by the Transcreation Framework for Community-engaged Behavioral Interventions to Reduce Health Disparities (Transcreation Framework), the overall purpose of this study is to determine the feasibility, acceptability, and preliminary efficacy of the proposed biobehavioral community-based and peer-led Black Breast Cancer Survivors Intervention (BBCSI) to improve QOL. To achieve this goal, I have assembled a strong mentorship team with complementary and relevant expertise to pursue the following specific aims:

Specific Aim 1: Develop a prototype of the BBCSI curriculum and assess satisfaction of the intervention. In partnership with two community-based organizations in Georgia and California; and guided by the Transcreation Framework, a prototype of the intervention and associated materials will be developed. Satisfaction of the content, materials, and intervention delivery procedures will be assessed through key informant interviews with Black breast cancer survivors (within two-years of diagnosis) and community interventionists.

Specific Aim 2: Determine the preliminary efficacy of the BBCSI. Using a one group, pre-post intervention design, we will assess improvements in QOL scores, health behaviors, and reduction of parabens in urine samples (markers of product use) of Black breast cancer survivors.

Specific Aim 3: Evaluate fidelity, feasibility, acceptability, barriers, and facilitators of the BBCSI. We will explore fidelity, feasibility, acceptability, barriers, and facilitators of intervention delivery through observation, surveys and key informant interviews with trained peer community interventionists, survivors, and community partner organizations.

The robust evidence of Black women's disproportionate exposure to carcinogenic chemicals that results in cancer-related disparities provides the impetus for this proposed intervention. I seek to fill a critical knowledge gap on developing, implementing, and analyzing community-based interventions. Dr. Teteh-Brook's strong mentorship team consists of leading experts in biological, and social influences on women's health (Glynn); randomized intervention design and implementation (Sun & Newton); clinical implications of intervention design for Black breast cancer survivors (Brewster); and environmental exposures assessments (Dodson). The PI's long-term career goal is to become an independent, community-based implementation researcher with a focus on environmental exposure behaviors related to Black identity and the proposed K01 application will help reach this goal. This K01 will produce training and findings to support an R01 to conduct a randomized trial of the BBCSI to establish efficacy and potential for dissemination/ implementation. Dr. Teteh-Brooks will use the findings from this proposed research to further refine and develop the trial design, infrastructure, and intervention delivery procedures.

ELIGIBILITY:
Inclusion Criteria:

Participants:

To be eligible to participate in this study, an individual must meet all the following criteria:

1. Adult women aged 18 years and older
2. Histologically confirmed stage 0-III breast cancer
3. No evidence of metastatic disease
4. Within four-years of diagnosis
5. Self-identify as Black
6. Able to communicate in English

Community Interventionists:

To be eligible to participate in this study, an individual must meet all the following criteria:

1. Adult women aged 18 years and older
2. Histologically confirmed stage 0-III breast cancer
3. No evidence of metastatic disease
4. Self-identify as Black
5. Able to communicate in English

Exclusion Criteria:

1. Men or woman below 18 years of age
2. Does not have a histologically confirmed breast cancer
3. There's evidence of metastatic disease
4. More than four-years of diagnosis
5. Does not self-identify as Black
6. Unable to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Time Frame: Through study completion; an average of 1 year
  Safety and Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Dede Teteh-Brooks, DRPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org